CLINICAL TRIAL: NCT00637403
Title: An Open-Label, Single-Dose Study to Assess the Effect of Renal Impairment on the Pharmacokinetic Characteristics, Safety, and Tolerability of Megestrol Acetate
Brief Title: Effect of Renal Impairment on the Pharmacokinetics, and Safety of Megestrol Acetate Concentrated Suspension
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty finding the required subject population
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: Covance (Industry); SFBC Anapharm (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 100.2.C.002
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: renal impairment; end stage renal disease; megestrol acetate; pharmacokinetics; hemodialysis; renal dialysis; kidney failure, chronic; renal insufficiency; Megace ES
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic | interventions — Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- I (Active Comparator): Megestrol acetate concentrated suspension in subjects with normal renal function
  Interventions: Drug: Megestrol acetate concentrated suspension 125 mg/mL
- II (Experimental): Megestrol acetate concentrated suspension in subjects with mild renal impairment
  Interventions: Drug: Megestrol acetate concentrated suspension 125 mg/mL
- III (Experimental): Megestrol acetate concentrated suspension in subjects with moderate renal impairment
  Interventions: Drug: Megestrol acetate concentrated suspension 125 mg/mL
- IV (Experimental): Megestrol acetate concentrated suspension in subjects with severe renal impairment
  Interventions: Drug: Megestrol acetate concentrated suspension 125 mg/mL
- V (Experimental): Megestrol acetate concentrated suspension in subjects with end stage renal disease
  Interventions: Drug: Megestrol acetate concentrated suspension 125 mg/mL

INTERVENTIONS:
Drug: Megestrol acetate concentrated suspension 125 mg/mL — Megestrol acetate concentrated suspension (125 mg/mL) administered orally for a total dose of 300 mg (2.4 mL x 125 mg/mL) in subjects with normal renal function (CLcr >80 mL/min)
  Other Names: Megace ES
  Arms: I
Drug: Megestrol acetate concentrated suspension 125 mg/mL — Megestrol acetate concentrated suspension (125 mg/mL) administered orally for a total dose of 300 mg (2.4 mL x 125 mg/mL) in subjects with mild renal impairment (CLcr 50 - 80 mL/min)
  Other Names: Megace ES
  Arms: II
Drug: Megestrol acetate concentrated suspension 125 mg/mL — Megestrol acetate concentrated suspension (125 mg/mL) administered orally for a total dose of 300 mg (2.4 mL x 125 mg/mL) in subjects with moderate renal impairment (CLcr 30 - <50 mL/min)
  Other Names: Megace ES
  Arms: III
Drug: Megestrol acetate concentrated suspension 125 mg/mL — Megestrol acetate concentrated suspension (125 mg/mL) administered orally for a total dose of 300 mg (2.4 mL x 125 mg/mL) in subjects with severe renal impairment (CLcr <30 mL/min and not on hemodialysis)
  Other Names: Megace ES
  Arms: IV
Drug: Megestrol acetate concentrated suspension 125 mg/mL — Megestrol acetate concentrated suspension (125 mg/mL) administered orally as 2 single doses of 300 mg (2.4 mL x 125 mg/mL) each in subjects with end stage renal disease undergoing hemodialysis. Washout period of 21 days between each dose
  Other Names: Megace ES
  Arms: V

SUMMARY:
To determine the pharmacokinetics and safety of megestrol acetate after a single oral 300 mg dose of megestrol acetate concentrated suspension in healthy subjects, and subjects with varying degrees of renal impairment

ELIGIBILITY:
Inclusion Criteria:

Healthy Subjects with Normal Renal Function

1. BMI ≥18 kg/m2 and ≤35 kg/m2
2. Females of child-bearing potential must use an adequate and reliable method of contraception. Postmenopausal females must be postmenopausal ≥1 year and have elevated serum FSH
3. Able to provide written informed consent
4. Normal renal function, defined as estimated creatinine clearance (CLcr) >80 mL/min at screening

Subjects with Mild, Moderate, or Severe Renal Impairment or ESRD

Meet inclusion criteria 1 through 3 for healthy subjects and the following criteria:

1. Renal impairment defined as creatinine clearance <80 mL/min as determined using the Cockroft-Gault formula. Subjects grouped according to degree of renal dysfunction: mild (CLcr = >50 and ≤80 mL/min), moderate (CLcr = >30 and ≤50 mL/min), or severe (CLcr = ≤30 mL/min)
2. Renal Impairment subjects must have evidence of stable renal impairment. Defined as having CLcr values within 25% of each other from 2 separately measured serum creatinine clearances using the Cockroft-Gault formula
3. ESRD subjects require hemodialysis for at least 3 months
4. Subjects with renal impairment or ESRD may have clinical laboratory test result deviations that are judged by the Investigator to be consistent with the renal condition of the subject or of no additional clinical significance for this study
5. Subjects with renal impairment or ESRD, must have stable underlying medical conditions for at least 90 days prior to the start of study participation
6. Renal impaired subjects may smoke up to 5 cigarettes per day

Exclusion Criteria:

Healthy Subjects with Normal Renal Function

1. Clinically significant (history of or active) cardiac, hepatic, renal, pulmonary, endocrine, neurological, infectious, gastrointestinal, hematologic, oncologic, or psychiatric disease that could put the subject at increased risk or could interfere with the objectives of the study
2. Presence of any screening laboratory values outside the range of normal values and deemed clinically significant by the Investigator
3. Use of a prescription drug within 14 days of study start, a non-prescription drug within 7 days of study start, or need of concomitant medication during the study
4. Use of any drugs or herbal products known to inhibit or induce liver enzymes involved in drug metabolism (CYP P450) within 30 days prior to 1st dose
5. History of allergic reaction or serum sickness to any drug or drug metabolites
6. Whole blood donation within 56 days prior to the first MA-CS dose or plasma donation within 7 days prior to the first MA-CS dose
7. Positive test for HIV antibody or hepatitis B surface antigen (positive HIV or hepatitis C antibody for ESRD subjects are acceptable)
8. Presence of drugs of abuse and/or alcohol
9. Participation in another investigational drug study within 30 days prior to the first MA-CS dose
10. History of recent drug abuse or alcohol addiction during past 2 years
11. Pregnant or breastfeeding
12. Consumption of grapefruit containing foods and beverages within 7 days prior to the first MA-CS dose
13. History of recurrent thromboembolic events, a thromboembolic event in past three months, or those still receiving long-term anticoagulation for thromboembolism

Subjects with Mild, Moderate, or Severe Renal Impairment or ESRD

Excluded if subjects meet exclusion criteria 4 through 13 for healthy subjects and the following criteria:

1. Unstable disease defined as concurrent medical conditions that change significantly within 90 days
2. Changes in concomitant medications within 14 days prior to first dose administration or expected changes during study participation
3. Subjects with a renal transplant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-05; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic blood samples | predose and serially through 264 hours post dose
Urine collection | Predose and serially through 264 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth C Lasseter, MD, Principal Investigator — SFBC International; Lynn D. Kramer, MD, Study Director — Par Pharmaceutical, Inc.
Locations (1):
- SFBC International, Miami, Florida, United States